CLINICAL TRIAL: NCT02514304
Title: Study of Risk Factors for Gastrointestinal Bleeding and of the Determinants of Non-fatal and Fatal Cardiovascular Events After Gastrointestinal Bleeding in Patients Receiving Antithrombotic Therapy for Cardiovascular Prevention
Brief Title: Study of the Risk Factors and Outcomes After Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); Bristol-Myers Squibb (Industry); Daiichi Sankyo (Industry)
Responsible Party: Principal Investigator, John Eikelboom, MD, Population Health Research Institute
Other Study IDs: INTERBLEED
Record Dates: First submitted 2015-07-29; First posted 2015-08-03 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Hemorrhage; Cardiovascular Diseases
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this multicenter, two component observational and standardized case-control study is to evaluate risk factors of gastrointestinal (GI) bleeding with a prospective 3-month and 12-month follow-up to examine outcomes and their possible causes.

DETAILED DESCRIPTION:
Antithrombotic therapies are effective for prevention of cardiovascular (CV) events but cause bleeding. Emerging evidence indicates that extra-cranial bleeding is just as important as myocardial infarction as a marker of risk for subsequent non-fatal and fatal CV events, but this issue has not been prospectively studied. If the association between bleeding and CV events is causal, prevention of bleeding, by targeting the risk factors, and prevention of the complications of bleeding, by targeting the causal pathways, could substantially reduce the burden of bleeding-related CV events. Progress in developing these approaches has been limited by a knowledge gap. Known risk factors do not fully explain bleeding risk and the investigators do not understand the mechanisms linking bleeding with adverse outcome and whether the association is causal.

One-half of bleeds that lead to CV events in patients receiving antithrombotic therapy arise in the GI tract. INTERBLEED plans to explore risk factors for GI bleeding, and outcomes after GI bleeding, in this well-circumscribed and important group using a case-control design with prospective 3 month and 12 month follow-up.

Specific objectives are to: (1) identify risk factors for GI bleeding and estimate their population attributable risk; (2) determine the risk of non-fatal and fatal CV events and functional outcomes after GI bleeding; and (3) explore the possible mechanisms linking GI bleeding with CV outcome.

INTERBLEED will recruit 2500 case-control pairs from centres in Argentina, Belgium, Brazil, China, Ireland and the Netherlands. Data will be collected on patient characteristics, medical history and, in cases, the work-up, management and outcomes after bleeding. The INTERBLEED results will help to develop new approaches to reducing the burden of bleeding-related CV events.

ELIGIBILITY:
Inclusion Criteria:

Cases

* Age ≥ 18 years at enrollment
* Written informed consent
* Confirmed cardiovascular disease
* Present to the hospital with GI tract bleed or develop GI tract bleed in hospital

Controls

* Age ≥ 18 years at enrollment
* Written informed consent
* Confirmed cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The community, inpatient/outpatient clinics (endoscopy clinics, stroke prevention clinics, cardiac/vascular clinics), emergency rooms
Sampling Method: Non-Probability Sample
Enrollment: 4745 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction, stroke or death | Up to one year

SECONDARY OUTCOMES:
Change in functional status from baseline to 3 months | 3 months
  Functional status measured by SAGE questionnaire
Change in functional status from baseline to 12 months | 12 months
  Functional status measured by SAGE questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: John Eikelboom, MD, Principal Investigator — Population Health Research Institute, McMaster University
Locations (1):
- Hamilton Health Sciences, PHRI, Hamilton, Ontario, Canada